CLINICAL TRIAL: NCT03439813
Title: Treating Anxiety After Stroke (TASK) Feasibility Randomized Controlled Trial
Brief Title: Treating Anxiety After Stroke (TASK)
Acronym: TASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/0253
Record Dates: First submitted 2018-01-16; First posted 2018-02-20 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Anxiety Disorders; Stroke; Transient Ischemic Attack
Keywords: stroke; transient ischemic attack; anxiety; psychotherapy
MeSH Terms: conditions — Anxiety Disorders; Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant receives one of the two TASK interventions. Both are considered active interventions for anxiety.
  Once started on the intervention participant may realise the type of intervention he has received, thus unblinding treatment allocation. Participants remain unaware of the contents of intervention given to the other group. Outcomes are self-completed by participants electronically to achieve assessor blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TASK-CBT (Experimental): Web and telephone-delivered cognitive behavioural therapy designed for anxiety after stroke and TIA. Six personalized telephone CBT sessions, one week apart by a trained and supervised medical professional using the TASK Therapist's Manual. Treatment website contains multimedia content to cover key CBT skills with weekly online tasks.
  Interventions: Behavioral: TASK-CBT
- TASK-Relax (Active Comparator): Web and telephone-supported relaxation therapy. Treatment website contains five relaxation exercises: i) audio- and visually-guided breathing exercise, ii) relaxing imagery and sounds, iii) music for relaxation, iv) audio-guided progressive muscle relaxation, and v) a selection of sounds of nature. Telephone instruction given and treatment website contains multimedia content to explain to participant how to practice relaxation regularly during the trial period.
  Interventions: Behavioral: TASK-Relax

INTERVENTIONS:
Behavioral: TASK-CBT — .Web and telephone-delivered cognitive behavioural therapy designed for anxiety after stroke and TIA. Six personalized telephone CBT sessions, one week apart by a trained and supervised medical professional using the TASK Therapist's Manual. Treatment website contains multimedia content to cover key CBT skills with weekly online tasks.
  Arms: TASK-CBT
Behavioral: TASK-Relax — Web and telephone-supported relaxation therapy. Treatment website contains five relaxation exercises: i) audio- and visually-guided breathing exercise, ii) relaxing imagery and sounds, iii) music for relaxation, iv) audio-guided progressive muscle relaxation, and v) a selection of sounds of nature. Telephone instruction given and treatment website contains multimedia content to explain to participant how to practice relaxation regularly during the trial period.
  Arms: TASK-Relax

SUMMARY:
The TASK (Treating Anxiety after StroKe) trial is a feasibility randomized controlled trial. It aims to evaluate the feasibility of i) web-enabled trial procedures, and ii) the TASK intervention in stroke and TIA patients

DETAILED DESCRIPTION:
Anxiety after stroke and transient ischaemic attack (TIA) is common. It is distressing and potentially debilitating. Currently, post-stoke psychological care is inadequate. There is no definitive evidence to guide treatment of anxiety post-stroke.

The TASK intervention is a centralized model for delivering personalised therapy for treating anxiety post-stroke using telephone and web-technology.

The TASK intervention includes:

* Treatment website and telephone support
* Learning ways to overcome anxiety after stroke/'mini-stroke'
* Relaxation techniques
* Weekly online tasks
* Therapeutic videos
* Text reminders and participant record card
* Useful links to stroke resources and websites

The investigators designed the TASK trial to be web-enabled, so that it can be conducted entirely remotely.

In the TASK feasibility randomized controlled trial, the investigators aim to evaluate the feasibility of:

i) web-enabled trial procedures: online recruitment, remote eligibility checking, electronic informed consent, online self-reported outcome surveys

ii) feasibility of the TASK intervention in stroke and TIA patients

This trial received a favourable opinion from the South East Scotland Research Ethics Committee (ref: 17/SS/0143)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above
2. A diagnosis of stroke (ischaemic, primary haemorrhagic) or TIA-probable, definite, or ocular
3. At least one month after being discharged to the community from clinic or hospital ward
4. Has anxiety symptoms

   a. at least one anxiety symptom should be present on the 6-item anxiety screening questions derived from GAD-7 and modified Fear Questionnaire(ref).
5. Have capacity to give informed consent
6. Able to communicate in English on the telephone
7. Can access the internet via a computer/ tablet/ smartphone
8. Residents within NHS Lothian regions (EH postcodes and FK1)

   Exclusion Criteria:
9. People already taking part in a clinical trial of treatment intended to improve psychosocial outcomes e.g. emotional distress, anxiety, depression, emotionalism, fatigue, social functioning, quality of life are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of web-enabled self-recruitment | At 20 weeks
  Number of participants recruited per month

SECONDARY OUTCOMES:
Unwanted effects arising from any of the TASK treatments | At 20 weeks
  % participants reported unwanted effects from allocated intervention
Feasibility of electronic informed consent form | At 20 weeks
  % of participants completed electronic informed consent
Feasibility of remote eligibility confirmation via electronic health records | At 20 weeks
  Time taken to confirm eligibility (in days): date of randomization - date of data request made
Feasibility of assessing intervention fidelity | At 20 weeks
  % of Therapist's record of content(s) delivered
Feasibility of online self-completed surveys at data collection time points | At 6 and 20 weeks
  % completed follow up surveys

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Chun, MRCP, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Midlothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chun HY, Carson AJ, Tsanas A, Dennis MS, Mead GE, Calabria C, Whiteley WN. Telemedicine Cognitive Behavioral Therapy for Anxiety After Stroke: Proof-of-Concept Randomized Controlled Trial. Stroke. 2020 Aug;51(8):2297-2306. doi: 10.1161/STROKEAHA.120.029042. Epub 2020 Jun 24. PMID 32576090
- [Derived] Chun HY, Carson AJ, Dennis MS, Mead GE, Whiteley WN. Treating anxiety after stroke (TASK): the feasibility phase of a novel web-enabled randomised controlled trial. Pilot Feasibility Stud. 2018 Aug 14;4:139. doi: 10.1186/s40814-018-0329-x. eCollection 2018. PMID 30128164

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT03439813/Prot_SAP_000.pdf